CLINICAL TRIAL: NCT01829308
Title: SBIRT Implementation for Adolescents in Urban Federally Qualified Health Centers
Acronym: ST@T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: RTI International (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01DA034258-01 (NIH); 1R01DA034258-01 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Alcohol-induced Disorders; Drug Users; Tobacco Use Disorder
Keywords: implementation; SBIRT; alcohol screening; drug screening; Brief Intervention; Referral to Treatment; adolescents; Federally Qualified Health Centers
MeSH Terms: conditions — Alcohol-Induced Disorders; Drug Misuse; Tobacco Use Disorder | interventions — General Practitioners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialist (Experimental): The brief interventions are delivered by behavioral health counselors.
  Interventions: Behavioral: The brief interventions are delivered by behavioral health counselors (Specialist)
- Generalist (Active Comparator): The brief interventions are delivered by the primary care provider.
  Interventions: Behavioral: The brief interventions are delivered by the primary care provider (Generalist)

INTERVENTIONS:
Behavioral: The brief interventions are delivered by behavioral health counselors (Specialist) — Behavioral Health Specialists perform the brief intervention. The screening and referral to treatment processes remain the same as with the Generalist condition.
  Arms: Specialist
Behavioral: The brief interventions are delivered by the primary care provider (Generalist) — Primary care providers perform the brief intervention. The screening and referral to treatment processes remain the same as with the Specialist condition.
  Arms: Generalist

SUMMARY:
The purpose of this study is to examine the implementation of two evidence-based intervention strategies of SBIRT (Generalist vs. Specialist) for adolescent alcohol, tobacco, other drug use, and HIV risk behaviors.

DETAILED DESCRIPTION:
Guided by Proctor's conceptual model of implementation research, the proposed study is a multi-site, cluster randomized trial to compare two principal strategies of SBIRT delivery within adolescent medicine. In the Generalist Strategy, the primary care provider delivers brief intervention (BI) for substance misuse. In the Specialist Strategy, BIs are delivered by behavioral health counselors. The 7 study sites, primary care clinics operated by a large, urban Federally Qualified Health Center in Baltimore, will be randomly assigned to implement SBIRT for adolescents using either the Generalist or Specialist strategies. Staff at each site will be trained in the assigned implementation strategy, and quarterly booster trainings will be provided during the implementation period. Implementation outcomes, including: penetration, costs/cost-effectiveness, acceptability, timeliness, fidelity/adherence, and patient satisfaction will be assessed during the 18-month-long implementation period using a complementary combination of administrative service encounter data, provider and patient surveys, and qualitative interviews. At the end of the active implementation period, all training and technical support activities will cease for 12 months in order to measure relative sustainability. The study will also examine the effectiveness of integrating HIV risk screening within an SBIRT model.

ELIGIBILITY:
Inclusion Criteria:

* clinic staff

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Penetration of BI within the Generalist and Specialist models | 12 months
  To examine the relative effectiveness of the Generalist condition v. the Specialist condition in terms of penetration of brief intervention (proportion of patients receiving brief intervention [BI] among those for whom a BI is indicated).

SECONDARY OUTCOMES:
Referral to Treatment | 12 months
  To examine the relative effectiveness of the Generalist condition v. the Specialist condition in terms of referral to specialty substance abuse treatment for those adolescents for whom such treatment is indicated.
Long term penetration of BI within the Generalist and Specialist models | 12 months
  To examine the long term relative effectiveness of the Generalist condition v. the Specialist condition in terms of penetration of brief intervention (proportion of patients receiving BI among those for whom a BI is indicated).
HIV sex-risk behavior screening as part of adolescent SBIRT process | 12 months
  To examine the feasibility and acceptability of integrating HIV risk behavior screening into adolescent primary care as part of an SBIRT program.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon G Mitchell, PhD, Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Total Health Care, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell SG, Gryczynski J, Schwartz RP, Kirk AS, Dusek K, Oros M, Hosler C, O'Grady KE, Brown BS. Adolescent SBIRT implementation: Generalist vs. Specialist models of service delivery in primary care. J Subst Abuse Treat. 2020 Apr;111:67-72. doi: 10.1016/j.jsat.2020.01.007. Epub 2020 Jan 20. PMID 32087839
- [Derived] Monico LB, Mitchell SG, Dusek K, Gryczynski J, Schwartz RP, Oros M, Hosler C, O'Grady KE, Brown BS. A Comparison of Screening Practices for Adolescents in Primary Care After Implementation of Screening, Brief Intervention, and Referral to Treatment. J Adolesc Health. 2019 Jul;65(1):46-50. doi: 10.1016/j.jadohealth.2018.12.005. Epub 2019 Mar 6. PMID 30850312